CLINICAL TRIAL: NCT07325825
Title: A Comparative Evaluation of the Effectiveness of Topical Licorice Extract Gel and Diode Laser 445 nm on Physiologic Gingival Pigmentation
Brief Title: Licorice Extract Gel Versus Diode Laser for Physiologic Gingival Pigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rania Mostafa Eissa, Master's degree researcher, department of Oral Medicine and Diagnosis, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RaniaEissa-Dent-1999
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Gingival Hyperpigmentation
Keywords: Gingival pigmentation; Diode laser; Licorice extract gel
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: intervention (control group): Diode laser 445 nm intervention (test group): topical licorice extract gel
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diode Laser Group (Active Comparator): Participants receive gingival depigmentation using a 445 nm diode laser.
  Interventions: Device: Diode Laser 445 nm
- Licorice Extract Gel Group (Experimental): Participants apply topical licorice extract gel to pigmented gingival areas three times daily.
  Interventions: Drug: Licorice Extract Gel

INTERVENTIONS:
Device: Diode Laser 445 nm — Gingival depigmentation performed using a diode laser with a wavelength of 445 nm in continuous wave mode at 1 W power.
  Arms: Diode Laser Group
Drug: Licorice Extract Gel — Topical licorice extract gel applied to pigmented gingival areas three times daily for one month, with continuation for a second and third month if required.
  Arms: Licorice Extract Gel Group

SUMMARY:
This randomized controlled clinical trial aims to compare the effectiveness of topical licorice extract gel and diode laser (445 nm) in the treatment of physiologic gingival pigmentation.

Twenty-four adult patients presenting with physiologic melanin pigmentation in the anterior esthetic zone of the maxillary or mandibular gingiva will be randomly allocated into two equal groups. One group will be treated with diode laser therapy, while the other group will receive topical licorice extract gel.

Clinical outcomes will be assessed using standardized gingival pigmentation indices and patient satisfaction questionnaires over a follow-up period of 36 weeks.

DETAILED DESCRIPTION:
This randomized controlled clinical trial will be conducted at the outpatient clinic of the Department of Oral Medicine, Periodontology, Oral Diagnosis and Oral Radiology, Faculty of Dentistry, Alexandria University, Egypt.

Eligible participants aged 18-50 years with physiologic gingival pigmentation will be randomly assigned into two groups. Group A will receive gingival depigmentation using a 445 nm diode laser, while Group B will receive topical licorice extract gel applied three times daily.

The intensity and distribution of gingival pigmentation will be evaluated using the Dummett-Gupta Oral Pigmentation Index (DOPI) and Gingival Pigmentation Index (GPI). Patient satisfaction will also be assessed. Clinical evaluations will be performed at baseline, 1 week, 4 weeks, 12 weeks and 36 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 to 50 years old) of either sex with physiologic melanin pigmentation in the anterior esthetic zone of the maxillary or mandibular gingiva.
* Systemically healthy individuals

Exclusion Criteria:

* Smokers
* Pregnant or lactating females
* Patients taking drugs associated with gingival pigmentation
* Patients with periodontal disease
* History of gingival depigmentation
* Known hypersensitivity to licorice extract
* Poor oral hygiene
* Presence of systemic diseases

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Change in gingival pigmentation intensity | Baseline, 1 week, 4 weeks, 12 weeks and 36 weeks
  Degree of gingival pigmentation assessed using the Dummett-Gupta Oral Pigmentation Index (DOPI; scores range from 0 to 3), with higher scores indicating increased pigmentation intensity.
Change in gingival pigmentation distribution | Baseline, 1 week, 4 weeks, 12 weeks and 36 weeks
  Gingival pigmentation distribution was assessed using the Gingival Pigmentation Index (GPI). The GPI is an ordinal scale ranging from 0 to 3, where 0 indicates absence of pigmentation and 3 indicates widespread gingival pigmentation. Higher scores represent greater extent of gingival pigment distribution (worse pigmentation).

SECONDARY OUTCOMES:
Participant Satisfaction | 3 months post-treatment
  Participant satisfaction was assessed using a study-specific questionnaire consisting of four questions evaluating perceived esthetic improvement, fulfillment of expectations, self-confidence related to smile appearance, and willingness to recommend the treatment. Responses were recorded as categorical (non-numerical) variables, and no numerical scale was calculated. Outcomes were analyzed descriptively, with more favorable responses indicating higher satisfaction.
Postoperative pain intensity (laser group only) | Immediately post-procedure, Day 1 and Day 7 postoperatively
  Postoperative pain intensity was assessed in the diode laser group only using the Visual Analog Scale (VAS; range 0-10), where 0 indicates no pain and 10 indicates the worst imaginable pain. This outcome was not applicable to the licorice extract gel group due to the non-invasive nature of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Oral Medicine and Diagnosis Clinic, Faculty of Dentistry, Alexandria University, Alexandria, Alexandria Governorate, Egypt